CLINICAL TRIAL: NCT03515967
Title: The Use of a Portable 3D Head Mounted Display With Integrated Eye Capture Technology (I-PAS) for the Objectification and Quantification of Signs and Symptoms Associated With the Diagnosis of Mild Traumatic Brain Injury (mTBI)
Brief Title: Testing Mild Traumatic Brain Injury (mTBI) in Diverse Athletic Groups
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit
Sponsor: University of Miami (Other)
Collaborators: Syneos Health (Other); Neurolign (Industry)
Responsible Party: Principal Investigator, Michael E. Hoffer, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20170209
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Brain Injuries, Traumatic
Keywords: concussion, mild traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Injured Athletes (Experimental): Athletes tested for mild traumatic brain injury (mTBI) after injury using the I-PAS goggles
  Interventions: Device: I-PAS Goggles
- Non-Injured Athletes (Active Comparator): Athletes tested for mild traumatic brain injury (mTBI) with no injury using the I-PAS goggles
  Interventions: Device: I-PAS Goggles

INTERVENTIONS:
Device: I-PAS Goggles — Portable, head-mounted display goggle system with integrated eye capture technology

SUMMARY:
Study will test the use of a short virtual reality driven goggle test as a means of detecting mTBI in a diverse group of athletes

ELIGIBILITY:
Inclusion Criteria:

1. Participants from 18 - 90 years of age who participate in all amateur athletics at the University of Miami to include all levels of sports whether National Collegiate Athletic Association (NCAA) or Club. Initial recruitment will include high intensity sports, including but not limited to Men's football, Men's and Women's Soccer, Men's and Women's Basketball, Men's and Women's Volleyball, Men's Baseball and Women's Softball, and Club sports to include Men's and Women's Lacrosse, Hockey, Rugby, and Field Hockey).
2. Participants from 18-90 years of age who are or have been engaged in Olympic level competitions as an active participant or team member.
3. Participants from 18-90 years of age who are engaged in professional sports as an active participant or formerly as a team member. Initial recruitment will include all motor sports, ice and field hockey, football, soccer, basketball, and rugby.

Exclusion Criteria:

1. History of brain injury resulting from a penetrating wound to the head.
2. Presence of aphasia and/or inability to give informed consent for participation
3. History of diagnosed neuropsychiatric disorders
4. Documented neurodegenerative disorders
5. Prior disorders of hearing and balance including:

   1. Meniere's disease
   2. Multiple sclerosis
   3. Vestibular neuritis
   4. Vestibular schwannoma
   5. Sudden sensorineural hearing loss
6. Cerebrovascular disorders
7. History of ear operation other than myringotomy tube in the past
8. Systemic disorders: e.g. chronic renal failure, cirrhosis of the liver, etc.
9. Presence of intra-cranial structural findings on imaging studies
10. Prisoners

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-04-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with mTBI | 45 months
  How many participants were detected to have mTBI following a sports-related injury

SECONDARY OUTCOMES:
Time to recover | 45 months
  Measuring the time (days) it takes for readiness to return to sports activity after sports-related injury for participants with a detected mTBI

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoffer, MD, Principal Investigator — University of Miami

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoffer ME, Balaban C, Szczupak M, Buskirk J, Snapp H, Crawford J, Wise S, Murphy S, Marshall K, Pelusso C, Knowles S, Kiderman A. The use of oculomotor, vestibular, and reaction time tests to assess mild traumatic brain injury (mTBI) over time. Laryngoscope Investig Otolaryngol. 2017 Apr 12;2(4):157-165. doi: 10.1002/lio2.74. eCollection 2017 Aug. PMID 28894835
- [Background] Balaban C, Hoffer ME, Szczupak M, Snapp H, Crawford J, Murphy S, Marshall K, Pelusso C, Knowles S, Kiderman A. Oculomotor, Vestibular, and Reaction Time Tests in Mild Traumatic Brain Injury. PLoS One. 2016 Sep 21;11(9):e0162168. doi: 10.1371/journal.pone.0162168. eCollection 2016. PMID 27654131